CLINICAL TRIAL: NCT01027559
Title: fMRI Studies of Emotional Circuitry in Major Depression: Treatment Changes
Brief Title: fMRI Study of Treatment Changes in Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 081348; R01MH064821 (NIH); 2R01MH064821-05A2 (NIH); DDTR A3-NSI (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2009-12-04; First posted 2009-12-08 (Estimated); Results first posted 2018-06-13 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Major Depression; Treatment
Keywords: Major Depression; Functional Magnetic Resonance Imaging; Emotional Circuitry; Cognitive Behavioral Therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Depressed Group: CBT (Active Comparator): Depressed participants randomized to receive Cognitive Behavioral Therapy (CBT) for treatment. A fMRI scan session will occur immediately prior to starting treatment, and their second fMRI scan will occur immediately following the completion of 12 weeks of therapy.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Healthy Control Group (No Intervention): Healthy controls will an fMRI scan session and their second fMRI scan session will occur approximately 12 weeks after.
- Depressed Group: SRT (Active Comparator): Depressed participants randomized to receive the antidepressant sertraline (SRT) for treatment. A fMRI scan session will occur immediately prior to starting treatment, and their second fMRI scan will occur immediately following the completion of 12 weeks of therapy.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — Depressed participants will be randomized to SRT or CBT treatment. For those in the SRT treatment condition, visits will involve dispensing medications, checking for side effects and administering the Hamilton Depression rating scale occurring at Day = 0 and on or about Day = 14, Day 28, Day 42, Day 56, Day 70 and Day 84. Depressed patients treated with SRT will titrate up to a maximum dose of 200 mg daily depending on tolerability and inadequate antidepressant response. Depressed subjects will start their SRT treatment once their first MRI and computer testing sessions are completed.
  Other Names: SRT
  Arms: Depressed Group: SRT
Behavioral: Cognitive Behavioral Therapy — Depressed participants will be randomized to SRT or CBT treatment. For those in the CBT treatment condition, visits for the CBT sessions will occur on or about Day = 3,Day = 7,Day = 10,Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, and Day 84. Visits to check for progress and administer the Hamilton Depression rating scale will occur at Day = 0 and on or about Day = 14, Day 28, Day 42, Day 56, Day 70 and Day 84. Depressed subjects will start their CBT treatment once their first MRI and computer testing sessions are completed.
  Other Names: CBT
  Arms: Depressed Group: CBT

SUMMARY:
The overall purposes of this research are to determine if Cognitive Behavioral Therapy (CBT) has the same healing effect on the brain for people with depression as traditional antidepressants do, and in comparison to healthy controls with no history of depression, to find out more about the causes of depression including differences in the extent of problems caused by depression. We hypothesize that CBT will have the same healing effect on the brain as antidepressants; that differences in brain activations created by the various tasks and genetic differences will help us understand differences in the type and severity of symptoms among the depressed subjects.

DETAILED DESCRIPTION:
The overall purposes of this research are to determine if Cognitive Behavioral Therapy (CBT) has the same healing effect on the brain for people with depression as traditional antidepressants do, to find out more about the causes of depression and why people differ in the extent of problems caused by depression, and to determine if certain differences in genes within populations are related to clinical symptoms.Genes we are examining for this study are COMT, BDNF, and 5-HTT long arm and short arm, as well as future genes that may be discovered to play a role in depression at a later time, and will be determined by examining saliva and blood samples. We are primarily studying depression by functional Magnetic Resonance Imaging (fMRI) which allows us to identify certain parts of the brain that show how the brain works in controlling negative feelings. Participants will be imaged while performing different tasks that are believed to activate emotional circuitry of the brain. Comparisons of activation patterns across these tasks will be used to characterize the cognitive mechanisms supported by different cortical regions, and to determine patterns of functional brain deficits in subjects with depression. Comparisons will also be made between changes that occur after treatment with an approved antidepressant and treatment with CBT.

ELIGIBILITY:
DEPRESSED GROUP:

Inclusion criteria:

1. Age 18-50
2. DSM-IV criteria for major depressive disorder (MDD)
3. Minimum Hamilton Rating Scale for Depression (HAMD) score > 18
4. Right handed
5. Capacity to give informed consent and follow study procedures
6. English speaking

Exclusion criteria:

1. Cannot give informed consent
2. Significant handicaps (e.g. visual or hearing loss, mental retardation) that would interfere with testing procedures
3. Does not speak English
4. Known primary neurological disorders
5. Any other factor that in the investigators judgment may affect patient safety or compliance (e.g. distance greater than 100 miles from clinic)
6. MRI contraindications e.g. foreign metallic implants, pacemaker
7. Known allergy or hypersensitivity to sertraline
8. Active suicidality
9. Severe or unstable medical illness or conditions or drugs that may cause depression
10. Any of the following diagnosed by DSM-IV: alcohol or substance abuse disorder, schizophrenia or other psychotic disorder, bipolar disorder, psychotic features of depression, current obsessive compulsive disorder (OCD) or panic disorder. In general, subjects with a history of other Axis I disorders prior to their depression will be excluded.
11. Current episode has failed to respond to adequate trials of two prior antidepressants for at least 6 weeks at therapeutic doses.
12. Treatment with sertraline for at least one month in past 3 months.
13. Current use of psychotropic prescription or nonprescription drugs or herbals (e.g. hypericum) except for limited use of certain hypnotics.
14. Current psychotherapy
15. Treatment with psychotropic drugs or drugs that affect the CNS such as beta-blockers or mood stabilizers.

CONTROL GROUP:

Inclusion criteria:

1. Age 18-50
2. No history of MDD
3. HAMD score < 7
4. Right handed
5. Capacity to give informed consent and follow study procedures
6. English speaking

Exclusion criteria:

1. Cannot give informed consent
2. Significant handicaps (e.g. visual or hearing loss, mental retardation) that would interfere with testing procedures
3. Does not speak English
4. Known primary neurological disorders
5. Any other factor that in the investigators judgment may affect patient safety or compliance (e.g. distance greater than 100 miles from clinic)
6. MRI contraindications e.g. foreign metallic implants, pacemaker
7. Severe or unstable medical illness or conditions or drugs that may cause depression
8. Any of the following diagnosed by DSM-IV: alcohol or substance abuse disorder, schizophrenia or other psychotic disorder, bipolar disorder, major depression, OCD or panic disorder.
9. Current use of psychotropic prescription or nonprescription drugs or herbals (e.g. hypericum) except for limited use of certain hypnotics.
10. Treatment with psychotropic drugs or drugs that affect the CNS such as beta-blockers or mood stabilizers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2009-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette I Sheline, MD, Principal Investigator — University of Pennsylvania; Charles Conway, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to being assigned to a group, 6 depressed participants dropped from the study before being assigned to treatment type.
Groups:
- Depressed Group: CBT: Depressed participants randomized to receive Cognitive Behavioral Therapy (CBT) for treatment. fMRI scan session occurs immediately prior to starting treatment, and a second fMRI scan will occur following 12 weeks of therapy.
  Cognitive Behavioral Therapy: Visits for the CBT sessions will occur on or about Day = 3,Day = 7,Day = 10,Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, and Day 84. Visits to check for progress and HAMD administration will occur at Day = 0 and on or about Day = 14, Day 28, Day 42, Day 56, Day 70 and Day 84.
- Depressed Group: Sertraline: Depressed participants randomized to receive sertraline (SRT) for treatment. fMRI scan session occurs immediately prior to starting treatment, and a second fMRI scan will occur following 12 weeks of therapy.
  Sertraline: Visits will involve dispensing medication, side effects assessment and HAMD administration occurring at Day = 0 and on or about Day = 14, Day 28, Day 42, Day 56, Day 70 and Day 84. Depressed patients treated with SRT will titrate up to a maximum dose of 200 mg daily depending on tolerability and inadequate antidepressant response.
Period: Overall Study
Arm/Group | Depressed Group: CBT | Healthy Control Group | Depressed Group: Sertraline
Started | 26 | 34 | 31
Completed | 20 | 26 | 22
Not Completed | 6 | 8 | 9

BASELINE CHARACTERISTICS:
Population: A total of 97 participants enrolled in the study (63 depressed and 34 controls). Of the 63 depressed participants enrolled in the study, 57 (26 CBT and 31 SRT) were assigned to a treatment group and completed at least some study-related activities. Six depressed participants dropped from the study before being assigned to treatment type.
Groups:
- Depressed Group: SRT: Depressed participants randomized to receive sertraline (SRT) for treatment. fMRI scan session occurs immediately prior to starting treatment, and a second fMRI scan will occur following 12 weeks of therapy.
  Sertraline: Visits will involve dispensing medication, side effects assessment and HAMD administration occurring at Day = 0 and on or about Day = 14, Day 28, Day 42, Day 56, Day 70 and Day 84. Depressed patients treated with SRT will titrate up to a maximum dose of 200 mg daily depending on tolerability and inadequate antidepressant response.
- Total: Total of all reporting groups
Arm/Group | Depressed Group: CBT | Depressed Group: SRT | Healthy Control Group | Total
Number analyzed (Participants) | 26 | 31 | 34 | 91
Age, Continuous [Mean (Full Range); unit: years] | 31.54 [18 to 48] | 33.29 [19 to 49] | 31.64 [18 to 48] | 32.16 [18 to 49]
Sex/Gender, Customized [Number; unit: participants]
  Female | 19 | 26 | 28 | 77
  Male | 7 | 5 | 5 | 19
Region of Enrollment [Number; unit: participants]
  United States | 26 | 31 | 34 | 91

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygen-level Dependent Activations During an Emotional Distractor Task Between fMRI Scans of Depressed Participants in the CBT Group and Control Participants.
Description: MRI imaging was completed on 50 participants (26 depressed who were randomized to the CBT group and 24 controls) for this analysis, including fMRI scans to evaluate regional brain activation in depression during an emotional distractor task. Image data from their baseline visit was processed and analyzed to show differences in blood oxygen-level dependent (BOLD) activations between depressed participants in the CBT group and control participants in a priori regions (amygdala and dorsolateral prefrontal cortex) during the task. The specified regions were masked on the images, and voxel-wise comparisons (ANOVAs) were performed to determine differences in activations between groups within these masked regions Positive values reflect a BOLD activation in that region; negative reflects a BOLD de-activation in that region.
Time Frame: baseline visit and 8-week follow-up
Population: fMRI data from a total of 26 depressed participants randomized to receive CBT and 24 control participants was analyzed. The primary aim was to compare depressed and control participants to evaluate regional brain activation during an emotional task, both at baseline and 8-week follow-up. The primary regions analyzed were the amygdala and DLPFC.
Measure: Mean (Standard Deviation); unit: Voxels
Groups:
- Depressed Group: Depressed participants randomized to receive Cognitive Behavioral Therapy (CBT) for treatment. A fMRI scan session will occur immediately prior to starting treatment, and their second fMRI scan will occur immediately following the completion of 12 weeks of therapy.
  Cognitive Behavioral Therapy: Depressed participants will be randomized to SRT or CBT treatment. For those in the CBT treatment condition, visits for the CBT sessions will occur on or about Day = 3,Day = 7,Day = 10,Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, and Day 84. Visits to check for progress and administer the Hamilton Depression rating scale will occur at Day = 0 and on or about Day = 14, Day 28, Day 42, Day 56, Day 70 and Day 84. Depressed subjects will start their CBT treatment once their first MRI and computer testing sessions are completed.
Arm/Group | Depressed Group | Healthy Control Group
Number analyzed (Participants) | 26 | 24
Voxels
  Amygdala - baseline | -18.74 (98.45) | 2.71 (141.09)
  DLPFC - baseline | 316.24 (199.83) | 411.2 (241.53)
  Amygdala - Time 2 | -16.82 (108.55) | -46.06 (97.10)
  DLPFC - Time 2 | 403.72 (248.02) | 421.51 (231.33)

2. Primary Outcome: Hamilton Depression Rating Scale Score at Baseline and 12 Weeks
Description: The patient was rated by a research team member among 17 dimensions/items pertaining to depression symptoms experienced over the last week. Each item is scored from 0 (=absent), up to 2 or 4 (depending on the item). The maximum total score on the assessment, indicating the most severe depression, would be 52. A total score of 0-7 is considered to be normal. Total scores of 20 or higher indicate moderate, severe, or very severe depression. A 50% or greater drop in Hamilton Depression Rating Scale signifies response to treatment.
Time Frame: Baseline and 12 weeks
Population: Numbers may differ from Participant Flow but these are the totals of those participants who had data at this time point for the Hamilton Depression Rating Scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Depressed Group: Sertraline: Depressed participants randomized to receive sertraline (SRT) for treatment. fMRI scan session occurs immediately prior to starting treatment, and a second fMRI scan will occur following 12 weeks of therapy.
  Sertraline: Visits will involve dispensing medication, side effects assessment and Hamilton Depression Rating Scale (HAMD) administration occurring at Day = 0 and on or about Day = 14, Day 28, Day 42, Day 56, Day 70 and Day 84. Depressed patients treated with SRT will titrate up to a maximum dose of 200 mg daily depending on tolerability and inadequate antidepressant response.
Arm/Group | Depressed Group: CBT | Healthy Control Group | Depressed Group: Sertraline
Number analyzed (Participants) | 18 | 15 | 14
units on a scale
  Baseline | 19.94 (5.23) | 1.38 (1.33) | 20.79 (3.98)
  Week 12 | 5.94 (6.08) | 1.07 (1.33) | 4.43 (5.37)

ADVERSE EVENTS:
Groups:
- Depressed Group: SSRI (Selective Serotonin Re-Uptake Inhibitor: Depressed participants randomized to receive setraline (SRT) for treatment. fMRI scan session occurs immediately prior to starting treatment, and a second fMRI scan will occur following 12 weeks of therapy.
  Sertraline: Visits will involve dispensing medication, side effects assessment and HAMD administration occurring at Day = 0 and on or about Day = 14, Day 28, Day 42, Day 56, Day 70 and Day 84. Depressed patients treated with SRT will titrate up to a maximum dose of 200 mg daily depending on tolerability and inadequate antidepressant response.
Arm/Group | Depressed Group: CBT | Healthy Control Group | Depressed Group: SSRI (Selective Serotonin Re-Uptake Inhibitor
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/34 | 0/31
Other Adverse Events (participants affected / at risk) | 7/26 | 2/34 | 21/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Depressed Group: CBT (N=26) | Healthy Control Group (N=34) | Depressed Group: SSRI (Selective Serotonin Re-Uptake Inhibitor (N=31)
Constipation (Gastrointestinal disorders) | 2 | 0 | 6
Sedation/Drowsiness (Nervous system disorders) | 4 | 0 | 17
Excitement/Weakness (Nervous system disorders) | 3 | 0 | 5
Headache (Nervous system disorders) | 3 | 0 | 12
Nausea/Vomitting (Gastrointestinal disorders) | 3 | 0 | 10
Stomach/Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 5
Irritability (Nervous system disorders) | 5 | 0 | 8
Muscle Twitching (Nervous system disorders) | 1 | 0 | 8
Tremor (Nervous system disorders) | 1 | 0 | 4
Decreased Appetite (Nervous system disorders) | 2 | 0 | 8
Increased Appetite (Nervous system disorders) | 2 | 0 | 5
Weight Gain (Nervous system disorders) | 2 | 0 | 5
Insomnia (Nervous system disorders) | 1 | 0 | 7
Dry Mouth (Immune system disorders) | 3 | 0 | 10
Decreased Libido (Nervous system disorders) | 2 | 0 | 7
Malaise (Immune system disorders) | 2 | 0 | 5
Impaired Mentation (Nervous system disorders) | 2 | 0 | 4
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Dizziness/Faintness (Ear and labyrinth disorders) | 1 | 0 | 8
Sexual Dysfunction (Nervous system disorders) | 0 | 0 | 6
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 5
Nasal Congestion (Immune system disorders) | 2 | 0 | 8
Excessive Sweating (Nervous system disorders) | 2 | 0 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 — Back pain/stiffness from taking part in the MRI scan
Chest Pain (Vascular disorders) | 1 | 0 | 2
Panic (Psychiatric disorders) | 0 | 0 | 2
Slurred Speech (Nervous system disorders) | 2 | 0 | 1
Difficulty Hearing/Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 3
Increased Libido (Vascular disorders) | 0 | 0 | 3
Syncope (Vascular disorders) | 0 | 0 | 2
Blurred Vision (Eye disorders) | 0 | 0 | 2
Increased Salivation (General disorders) | 0 | 0 | 2
Tachycardia/Palpitations (Cardiac disorders) | 0 | 0 | 2
Menstrual Irregularity (Reproductive system and breast disorders) | 0 | 0 | 2
Weight Loss (General disorders) | 0 | 0 | 3
Abnormal Muscle Tone/Movements (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No